CLINICAL TRIAL: NCT00408902
Title: Phase II Study of MLN518 in Patients With Metastatic Clear Cell Renal Cell Carcinoma
Brief Title: Tandutinib in Treating Patients Who Have Undergone Surgery for Metastatic Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03014; CASE 10805; CDR0000518799; U01CA062502 (NIH)
Record Dates: First submitted 2006-12-06; First posted 2006-12-07 (Estimated); Results first posted 2015-02-04 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-10

CONDITIONS: Clear Cell Renal Cell Carcinoma; Recurrent Renal Cell Cancer; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — tandutinib

ARMS (1):
- TandutinibTreatment (Experimental): Patients receive oral tandutinib 500 mg twice daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: tandutinib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: tandutinib — Given orally, 500 mg bid daily
  Other Names: CT53518; MLN518
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well tandutinib works in treating patients who have undergone surgery for metastatic kidney cancer. Tandutinib may stop the growth of kidney cancer by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving tandutinib after surgery may kill any tumor cells that remain after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the overall efficacy of MLN518 in patients with metastatic clear cell renal carcinoma.

SECONDARY OBJECTIVES:

I. To evaluate the effect of MLN518 on progression-free survival and overall survival in patients with metastatic clear cell renal carcinoma.

II. To evaluate the toxicity of MLN518 in patients with metastatic clear cell renal carcinoma.

III. To evaluate the effects of MLN518 on serum VEGF-A, VEGF-R2, PIGF, and PDGF levels of patients with metastatic renal cell carcinoma receiving MLN518.

IV. To determine the VHL gene status, methylation, and pVHL in archived material from the primary nephrectomy specimen of patients receiving MLN518.

V. To evaluate tumor blood flow and vessel permeability based on functional imaging with dynamic contrast enhanced magnetic resonance imaging (dceMRI) in metastatic renal cell carcinoma patients treated with MLN518.

OUTLINE: This is an open-label, nonrandomized study.

Patients receive oral tandutinib twice daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed RCC of clear cell histology; subjects must have a component of conventional clear cell RCC with or without sarcomatoid features
* Patients must have evidence of metastatic disease and must have had a cytoreductive nephrectomy at least 28 days prior to first day of treatment
* Archival tissue from nephrectomy must be available for correlative studies
* Patients must have measurable disease, defined by RECIST criteria
* Patients must have received at least one prior FDA approved therapy for metastatic renal cell carcinoma with either Sutent, or Nexavar, and may have received up to three prior systemic therapies for metastatic disease; prior cytokine therapy is also permitted
* Prior systemic therapy with other antiangiogenic agents such as Thalidomide, Bevacizumab, or AG013736 is permitted
* Patients must have a life expectancy of >= 3 months
* Patients must have an ECOG performance status of 0-1 (Karnofsky >= 70%)
* Patients must be at least 4 weeks from radiation therapy and recovered from all related toxicity
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 8.5 g/dl
* Total Bilirubin =< 1.5 X institutional upper limit of normal
* AST (SGOT)/ALT (SGPT) =< 3.5 X institutional upper limit of normal
* Alkaline phosphatase =< 2.5 ULN (=< 10 x ULN in presence of bone metastasis)
* Serum calcium of =< 12 mg/dl
* Creatinine =< 1.5 X institutional upper limit of normal
* INR =< 1.5, except for subjects receiving warfarin therapy; for subjects who are receiving warfarin for prophylaxis or treatment of thrombosis, INR values should be carefully monitored while patients are on study
* Electrocardiogram (12-lead) with cQTC < 500 msec using the Bazett's formula
* Absence of significant effusions and/or ascites
* No major surgery requiring general anesthesia within the past 28 days
* Patients may not have had brain metastasis
* Eligibility of patients receiving any medications or substances known to affect or with the potential to affect the activity or pharmacokinetics of MLN518 will be determined following review of their case by the Principal Investigator; because MLN518 is a substrate of the P-glycoprotein (P-gp) drug efflux pump, co- administration of agents that inhibit or induce this mechanism may alter exposure to MLN518
* The effects of MLN518 on the developing human fetus at the recommended therapeutic dose are unknown; for this reason and because receptor tyrosine kinase inhibitors are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; sexually active patients must continue to use contraception for three months after completion of study therapy
* All patients must be informed of the investigational nature of this study and must provide written informed consent in accordance with institutional and federal guidelines; a copy of the informed consent document signed by the patient must be given to the patient

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents
* Patients may not be co-medicated with an agent that causes QTc prolongation
* Patients with a mean QTc > 500 msec using the Bazett's formula taken from the screening electrocardiogram or history of familial long QT syndrome are ineligible
* Left ventricular ejection fraction (LVEF) < 40%
* Myocardial infarction within 6 months of enrollment or New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* Ongoing vomiting, or nausea >= grade 2 (NCI CTCAE v3.0)
* Patients with any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow pills or absorb oral medications are excluded
* Known or suspected primary muscular or neuromuscular disease (e.g., muscular dystrophy, myasthenia gravis)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MLN518 such as Tarceva™, Iressa® and Cardura® XL
* Patients with any CNS metastases or uncontrolled seizure disorder
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infections or psychiatric illness/social situations that would limit compliance with study requirements
* Any malignancy other than a renal cell carcinoma, with the following exceptions:

  * Basal or squamous cell carcinomas of the skin
  * Carcinoma in-situ of the uterine cervix
  * Any malignancy treated with curative intent and in complete remission for > 3 years
* Patients with organ allografts
* Patients with non-clear cell carcinoma i.e., papillary, collecting duct, or chromophobe
* Pregnant women are excluded from this study because MLN518 is a receptor tyrosine kinase inhibitor with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with MLN518, breastfeeding should be discontinued if the mother is treated with MLN518
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with MLN518; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Inability to comply with study and/or follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-11; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Garcia, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from Cleveland Clinic between November 2006 and August 2007.
Period: Overall Study
Arm/Group | TandutinibTreatment
Started | 10
Completed | 0
Not Completed | 10
Not completed — Lack of Efficacy | 7
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Arm/Group | TandutinibTreatment
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Overall Efficacy, Taking Into Account Both Objective Response and Meaningful Reductions in Tumor Burden That do Not Meet the RECIST Criteria for PR or CR (e.g., 5-30% Reduction in RECIST Defined Tumor Burden)
Description: The number of patients that reach complete response (CR)defined as the disappearance of all target lesions or partial response (PR)defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD.
Time Frame: Up to 4 weeks after completion of study treatment
Population: Intent to treat
Measure: Number; unit: participants
Groups:
- TandutinibTreatment: Patients receive oral tandutinib twice daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | TandutinibTreatment
Number analyzed (Participants) | 10
participants
  Complete Response (CR) | 0
  Partial Response (PR) | 0

2. Secondary Outcome: Overall Survival
Description: Estimated using the method of Kaplan and Meier.
Time Frame: Followed until progression or death for approximately 3 years
Population: Data was not collected as study closed prior to time period for analysis.
Arm/Group | TandutinibTreatment
Number analyzed (Participants) | 0

3. Secondary Outcome: Progression-free Survival
Description: Estimated time to progression using the method of Kaplan and Meier.
Time Frame: Up to 4 weeks after completion of study treatment
Population: Intent to treat
Measure: Median (Full Range); unit: months
Arm/Group | TandutinibTreatment
Number analyzed (Participants) | 10
months | 1.5 [0.9 to 2.1]

ADVERSE EVENTS:
Time Frame: Adverse events were collected while patients were on treatment and 4 weeks after treatment, up to 12 weeks.
Groups:
- TandutinibTreatment: Patients receive oral tandutinib twice daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  tandutinib: Given orally
  laboratory biomarker analysis: Correlative studies
Arm/Group | TandutinibTreatment
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TandutinibTreatment (N=10)
Fatigue (General disorders) | 3
Hemolysis (Blood and lymphatic system disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TandutinibTreatment (N=10)
Anorexia (Metabolism and nutrition disorders) | 1
Blood Urea Nitrogen (Metabolism and nutrition disorders) | 1
Chest pain (non-cardiac and non-pleuritic) (Musculoskeletal and connective tissue disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Creatinine (Investigations) | 3
Depression (Psychiatric disorders) | 1
Diarrhea patients without colostomy (Gastrointestinal disorders) | 8
Dizziness/lightheadedness (Nervous system disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3
Edema (Vascular disorders) | 5
Fatigue (lethargy, malaise, asthenia) (General disorders) | 4
Gastrointestinal-distention/bloating (Gastrointestinal disorders) | 2
Hearing w/o monitoring (Ear and labyrinth disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 7
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Investigations) | 1
Hypothyroidism (Endocrine disorders) | 1
Hypouricemia (Renal and urinary disorders) | 1
Insomnia (Psychiatric disorders) | 2
Lymphopenia (Blood and lymphatic system disorders) | 2
Mood alteration-anxiety, agitation (Psychiatric disorders) | 1
Muscle weakness (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 2
Nausea (Gastrointestinal disorders) | 7
Pain (Musculoskeletal and connective tissue disorders) | 3
Palpitations (Cardiac disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Prolonged QTc interval (QTc > 0.48 seconds) (Investigations) | 2
Protein (Renal and urinary disorders) | 1
Retroperitoneal hemorrhage (Gastrointestinal disorders) | 1
Rigors, chills (General disorders) | 3
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 1
Tearing (watery eyes) (Eye disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Vision-blurred vision (Eye disorders) | 1
Voice changes/stridor/larynx (e.g., hoarseness, loss of voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 7
Weight gain (Metabolism and nutrition disorders) | 1
Weight loss (Metabolism and nutrition disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1

LIMITATIONS AND CAVEATS:
Principal Investigator closed this study due to lack of response and toxicities of drug, therefore overall survival analysis was not done.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less